CLINICAL TRIAL: NCT03029156
Title: Effectiveness of the Aeroneb Compared to a Jet Nebulizer Fort the Delivery of Bronchodilator Therapy of Acute Severe Asthma
Brief Title: Effectiveness of the Aeroneb in Acute Severe Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 11643
Record Dates: First submitted 2016-07-18; First posted 2017-01-24 (Estimated); Results first posted 2023-05-19 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Asthma Exacerbation
Keywords: Asthma; Aeroneb; Aerogen; Bronchodilator
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Small volume jet nebulizer (Active Comparator): Administration of bronchodilator through small volume jet nebulizer. The nebulized solution contains ipratropium / albuterol.
  Interventions: Device: Small volume jet nebulizer
- Aeroneb nebulizer (Experimental): Administration of bronchodilator via Aeroneb nebulizer. The nebulized solution contains ipratropium / albuterol.
  Interventions: Device: Aeroneb nebulizer

INTERVENTIONS:
Device: Aeroneb nebulizer — The Aeroneb Nebulizer System is a portable medical device for single patient use that is intended to aerosolize physician-prescribed solutions for inhalation to patients on and off ventilation.
  The Aeroneb Adapter is an accessory specific to the Aeroneb Nebulizer. It facilitates intermittent and continuous nebulization and optional supply of supplemental oxygen to adult patients in hospital use environments via a mouthpiece or aerosol mask. The Aeroneb Nebulizer System and Adapter are FDA approved devices for nebulizing solutions including bronchodilators (albuterol and ipratropium).
  Other Names: Vibrating mesh nebulizer
  Arms: Aeroneb nebulizer
Device: Small volume jet nebulizer — The bronchodilators will be administered via small volume jet nebulizer
  Arms: Small volume jet nebulizer

SUMMARY:
Background: The bronchodilator therapy is an essential component of the management of asthma exacerbation. The delivery of bronchodilators to the lungs in asthma exacerbations is usually achieved through nebulization (creating small particles to be inhaled). The commonly used nebulizer device is a small volume jet nebulizer which has not been consistently reliable in delivering bronchodilator therapy. The Aeroneb nebulizer device is a FDA approved device which produces consistently respirable sized particles which could potentially result in better bronchodilator effect than the standard jet nebulizer.

Aim: To study whether the Aeroneb nebulizer is more effective than a small volume jet nebulizer in delivering bronchodilators during a severe asthma exacerbation.

Experimental design: Patients will be randomized (like a flip of a coin) to receive bronchodilator therapy as per the emergency room protocol either via small volume jet nebulizer or Aeroneb nebulizer.

Subjects: Adult patients between age of 18 and 55 years who present to the emergency room with severe asthma exacerbation with peak expiratory flow rate <50% of predicted.

Study procedure: When enrolled in the study and after randomization, we will then collect data that is standard for the hospital like heart rate, blood pressure and breathing indices and also some non-routine things like some scoring scales for shortness of breath and serial measurements of peak expiratory flow rate. We anticipate that the Aeroneb device will be more effective in delivering bronchodilator medication and thus more effective in managing asthma exacerbations.

DETAILED DESCRIPTION:
* Patients presenting with acute severe asthma exacerbations to the emergency room will be screened by the PI, co-investigator or research coordinator to determine their eligibility based on the inclusion and exclusion criteria.
* Clinically indicated treatment must not be delayed for a research-related reason so patients will still be eligible for enrollment after receiving initial bronchodilator therapy as long as their PEFR remains <50% of predicted and enrollment occurs within 90 minutes of the ER arrival time.
* The initial part of the consent process will cover the essential elements of the informed consent in a concise manner to ensure a timely process
* Eligible patients will be randomized using the concealed envelope method to either the intervention arm or the control arm. The randomization should take place within 90 minutes of ER arrival, however, every effort will be made to enroll the patient as soon as possible; patients will be enrolled as long as their PEFR is less than 50% of predicted regardless of the number of bronchodilator treatments they received prior to randomization.
* The assignment will be blinded to the recording investigator and the treating physician but not to the patient or the nurse or respiratory therapist who is administering the nebulization. In order to avoid any delay in administering the treatments, the sets of Aeroneb nebulizer and small volume jet nebulizer will be stored in identical boxes and will be readily available in the ER.

In order to blind the treating physician and the recording investigator, a sign "treatment in progress" will be displayed at the outdoor of the ER room when the patient is getting the bronchodilator treatment. The nebulizer devices will be placed in the box between the bronchodilator treatment sessions. The physician and the recording investigator will be asked if possible to see the patients only when the sign is taken off the outdoor.

* Once assigned, all the bronchodilator treatments in the ER will be administered using the nebulizer device assigned to that patient.
* The Peak flow and FEV1 will be measured using Spirometer (micro I). Both values will be obtained through the same exhalation maneuver.
* Patient will be treated and managed according to the asthma ER adult protocol or as directed by the ER physician who is in charge of patient's care
* After the study procedures have been performed and the subject is determined to be in stable condition and have the capacity to make medical decisions, the investigator will approach the subject again and review all the elements of the ICF again with the subject. The collected data will be used only if the subject signs both parts of the informed consent.
* Within two weeks of the subject participation, the research team will conduct a phone interview with the subject to obtain their feedback on the study procedures and mainly on the informed consent process. The phone interview questionnaire is included in the supplement

ELIGIBILITY:
Inclusion Criteria:

* Acute asthma exacerbations presenting to the emergency room
* Peak expiratory flow rate at presentation <40% of predicted
* Enrolment within 90 minutes of the arrival to the ER
* Age 18-55 years old

Exclusion Criteria:

* History of chronic obstructive pulmonary disease
* Clinical evidence to suggest a non-asthmatic cause of bronchospasm as determined by the treating physician
* Clinical evidence of acute coronary syndrome
* Respiratory failure requiring mechanical ventilation either invasive or non-invasive
* Tachyarrhythmia other than sinus
* Agitated or uncooperative
* Inability to provide informed consent

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas S Hill, MD, Principal Investigator — Tufts Medical Center
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McFadden ER Jr. Acute severe asthma. Am J Respir Crit Care Med. 2003 Oct 1;168(7):740-59. doi: 10.1164/rccm.200208-902SO. PMID 14522812
- [Background] National Asthma Education and Prevention Program. Expert Panel Report 3 (EPR-3): Guidelines for the Diagnosis and Management of Asthma-Summary Report 2007. J Allergy Clin Immunol. 2007 Nov;120(5 Suppl):S94-138. doi: 10.1016/j.jaci.2007.09.043. PMID 17983880
- [Background] Rodrigo G, Rodrigo C. A new index for early prediction of hospitalization in patients with acute asthma. Am J Emerg Med. 1997 Jan;15(1):8-13. doi: 10.1016/s0735-6757(97)90039-5. PMID 9002561
- [Background] Rodrigo G, Rodrigo C. Early prediction of poor response in acute asthma patients in the emergency department. Chest. 1998 Oct;114(4):1016-21. doi: 10.1378/chest.114.4.1016. PMID 9792570
- [Background] Piovesan DM, Menegotto DM, Kang S, Franciscatto E, Millan T, Hoffmann C, Pasin LR, Fischer J, Barreto SS, Dalcin Pde T. Early prognosis of acute asthma in the emergency room. J Bras Pneumol. 2006 Jan-Feb;32(1):1-9. doi: 10.1590/s1806-37132006000100004. English, Portuguese. PMID 17273562
- [Background] Ari A, Atalay OT, Harwood R, Sheard MM, Aljamhan EA, Fink JB. Influence of nebulizer type, position, and bias flow on aerosol drug delivery in simulated pediatric and adult lung models during mechanical ventilation. Respir Care. 2010 Jul;55(7):845-51. PMID 20587095
- [Background] Galindo-Filho VC, Ramos ME, Rattes CS, Barbosa AK, Brandao DC, Brandao SC, Fink JB, de Andrade AD. Radioaerosol Pulmonary Deposition Using Mesh and Jet Nebulizers During Noninvasive Ventilation in Healthy Subjects. Respir Care. 2015 Sep;60(9):1238-46. doi: 10.4187/respcare.03667. Epub 2015 Jun 23. PMID 26106207
- [Background] Alvine GF, Rodgers P, Fitzsimmons KM, Ahrens RC. Disposable jet nebulizers. How reliable are they? Chest. 1992 Feb;101(2):316-9. doi: 10.1378/chest.101.2.316. PMID 1735247
- [Background] Borg G. Perceived exertion as an indicator of somatic stress. Scand J Rehabil Med. 1970;2(2):92-8. No abstract available. PMID 5523831
- [Background] Patrick W, Webster K, Ludwig L, Roberts D, Wiebe P, Younes M. Noninvasive positive-pressure ventilation in acute respiratory distress without prior chronic respiratory failure. Am J Respir Crit Care Med. 1996 Mar;153(3):1005-11. doi: 10.1164/ajrccm.153.3.8630538.

RESULTS

PARTICIPANT FLOW:
Groups:
- Aeroneb Nebulizer: Administration of bronchodilator via Aeroneb nebulizer. The nebulized solution contains ipratropium / albuterol.
  The Aeroneb Nebulizer System is a portable medical device for single patient use that is intended to aerosolize physician-prescribed solutions for inhalation to patients on and off ventilation.
  The Aeroneb Adapter is an accessory specific to the Aeroneb Nebulizer. It facilitates intermittent and continuous nebulization and optional supply of supplemental oxygen to adult patients in hospital use environments via a mouthpiece or aerosol mask. The Aeroneb Nebulizer System and Adapter are FDA approved devices for nebulizing solutions including bronchodilators (albuterol and ipratropium).
Period: Overall Study
Arm/Group | Small Volume Jet Nebulizer | Aeroneb Nebulizer
Started | 15 | 16
Completed | 15 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Small Volume Jet Nebulizer | Aeroneb Nebulizer | Total
Number analyzed (Participants) | 15 | 16 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.4 (8.46) | 39.9 (9.05) | 36 (8.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 10 | 18
  Male | 7 | 6 | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: African American | 4 | 7 | 11
  Race/Ethnicity: Asian | 2 | 0 | 2
  Race/Ethnicity: Hispanic | 2 | 2 | 4
  Race/Ethnicity: White | 7 | 7 | 14

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in Mean of Peak Expiratory Flow Rate (PEFR) Percentage of Predicted Baseline at 30 Minutes After the Initial Bronchodilator Treatment
Description: Peak expiratory flow rate is the maximum flow rate generated during a forceful exhalation, starting from full inspiration.
Time Frame: 30 minutes
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Small Volume Jet Nebulizer | Aeroneb Nebulizer
Number analyzed (Participants) | 15 | 16
percent change | 18.1 (18.01) | 12.9 (13.36)

2. Secondary Outcome: Percentage Change in the PEFR Percentage of Predicted Baseline to Disposition
Description: Change in the PEFR percent predicted from the initial bronchodilator treatment in the Aeroneb group compared to the small volume jet nebulizer group.
Time Frame: Initial bronchodilator treatment to disposition, an average of 4 hours
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Small Volume Jet Nebulizer | Aeroneb Nebulizer
Number analyzed (Participants) | 15 | 16
percent change | 23.3 (15.15) | 14.4 (14.04)

3. Secondary Outcome: Percentage Change in the Forced Expiratory Volume (FEV1) Percentage of Predicted Baseline to Disposition
Description: Forced expiratory volume refers to the volume of air that an individual can exhale during a forced breath in 1 second.
Time Frame: initial bronchodilator treatment to disposition, an average of 4 hours
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Small Volume Jet Nebulizer | Aeroneb Nebulizer
Number analyzed (Participants) | 15 | 16
percent change | 17.1 (13.05) | 8.0 (8.08)

4. Secondary Outcome: Change in the Borg-Dyspnea Score From Baseline to Disposition
Description: The Borg-Dyspnea score measures an individual's effort, exertion, breathlessness and fatigue during physical work. This scale ranges from 6-20 with 6 representing no exertion at all and 20 representing maximal exertion.
Time Frame: initial bronchodilator treatment to disposition, an average of 4 hours
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Small Volume Jet Nebulizer | Aeroneb Nebulizer
Number analyzed (Participants) | 15 | 16
score on a scale | 2.44 (0.12) | 3.15 (1.01)

5. Secondary Outcome: Change in Heart Rate Baseline to Disposition
Description: Change in the heart rate at baseline after the initial bronchodilator treatment in the Aeroneb group compared to the small volume jet nebulizer group.
Time Frame: The initial bronchodilator treatment to to disposition, an average of 4 hours
Measure: Mean (Standard Deviation); unit: Change in heart rate (beats/min)
Arm/Group | Small Volume Jet Nebulizer | Aeroneb Nebulizer
Number analyzed (Participants) | 15 | 16
Change in heart rate (beats/min) | 1 (3) | 1 (5)

6. Secondary Outcome: Length of Stay in the ER
Description: Total length from admission to discharge.
Time Frame: Length of stay in the ER - up to one day
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Small Volume Jet Nebulizer | Aeroneb Nebulizer
Number analyzed (Participants) | 15 | 16
minutes | 272.3 (123.74) | 245.3 (139.36)

7. Secondary Outcome: Percentage of Patients Requiring Hospitalization
Description: Total amount of patients requiring hospitalization after ER admission.
Time Frame: Length of stay in the ER - up to one day
Measure: Count of Participants; unit: Participants
Arm/Group | Small Volume Jet Nebulizer | Aeroneb Nebulizer
Number analyzed (Participants) | 15 | 16
Participants | 4 | 6

8. Secondary Outcome: The Total Dose of Albuterol Used in Each Group During ED Stay
Description: Albuterol is used to prevent and treat difficulty breathing, wheezing, shortness of breath, coughing, and chest tightness caused by lung diseases such as asthma and chronic obstructive pulmonary disease.
Time Frame: Length of stay in the ER - up to one day
Measure: Mean (Standard Deviation); unit: dosage (mg)
Arm/Group | Small Volume Jet Nebulizer | Aeroneb Nebulizer
Number analyzed (Participants) | 15 | 16
dosage (mg) | 6.3 (2.97) | 7.2 (4.07)

9. Other Pre Specified Outcome: The Total Dose of Ipratropium Used in Each Group During ED Stay
Description: Ipratropium is used to prevent wheezing, shortness of breath, coughing and chest tightness in people with chronic obstructive pulmonary disease, chronic bronchitis, and emphysema. It is a bronchodilator which relaxes and opens the air passages to the lungs to make breathing easier.
Time Frame: Length of stay in the ER - up to one day
Measure: Mean (Standard Deviation); unit: dosage (mg)
Arm/Group | Small Volume Jet Nebulizer | Aeroneb Nebulizer
Number analyzed (Participants) | 15 | 16
dosage (mg) | 1 (0.44) | 1.1 (0.56)

ADVERSE EVENTS:
Time Frame: Adverse events data was collected for 2 years, the duration of the study.
Arm/Group | Small Volume Jet Nebulizer | Aeroneb Nebulizer
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/16
Other Adverse Events (participants affected / at risk) | 0/15 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-20): https://cdn.clinicaltrials.gov/large-docs/56/NCT03029156/Prot_SAP_000.pdf